CLINICAL TRIAL: NCT05472350
Title: Efficacy and Safety of Perioperative Use of Breztri Aerosphere to Relieve Cough After Lobectomy: A Prospective, Randomized, Placebo-controlled Single Center Trial
Brief Title: Efficacy and Safety of Perioperative Use of Breztri Aerosphere to Relieve Cough After Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, Director, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAH20220717
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer, Nonsmall Cell; Perioperative; Cough; Drug Effect; Drug Toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cough; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breztri Aerosphere Group (Experimental): Participants will receive Breztri Aerosphere twice a day from 3 days before surgery to 14 days after surgery
  Interventions: Drug: Breztri Aerosphere
- Placebo Group (Placebo Comparator): Participants will receive 0.9% normal saline twice a day from 3 days before surgery to 14 days after surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Breztri Aerosphere — Breztri Aerosphere is used to control and prevent symptoms (such as wheezing and shortness of breath) caused by ongoing lung disease (chronic obstructive pulmonary disease-COPD, which includes chronic bronchitis and emphysema).
  Arms: Breztri Aerosphere Group
Other: Placebo — placebo is 0.9% normal saline
  Arms: Placebo Group

SUMMARY:
Cough after lobectomy is common. The prevention and treatment of cough after lobectomy is not standardized. Breztri Aerosphere is often used to relieve cough. Therefore, we conduct a single center placebo-controlled study to evaluate the efficacy and safety of perioperative use of Breztri Aerosphere in relieving cough after lobectomy.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized, controlled clinical trial to understand the efficacy and safety of perioperative use of Breztri in relieving cough after lobectomy. This study plans to include 128 subjects from the Department of Thoracic Surgery of the First Affiliated Hospital of Guangzhou Medical University. Participants will be randomly divided into according Breztri group and placebo group to the ratio of 1:1. Participants in Placebo group will receive 0.9% normal saline for 3 days before operation and 14 days after operation (n=64). Participants in Breztri group will receive Breztri for 3 days before operation and 14 days after operation (n=64). All patients will undergo screening and baseline visits. After sugery, they will be followed up for 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this research and abide by the research regulations, understand and comply with and cooperate with the corresponding inspections, comply with the follow-up plan, and voluntarily sign the written informed consent.
2. Outpatients, 18 years old ≤ age ≤ 70 years old, preoperative examination of cardiopulmonary function can tolerate surgery.
3. Patients planning to undergo lobectomy.
4. No obvious cough before surgery.

Exclusion Criteria:

1. Participated in other interventional clinical trials 90 days before enrollment
2. Pregnant and lactating women (budigrafo is not recommended during pregnancy and lactation)
3. Patients with obvious cough before surgery (which affects the evaluation of drug effect)
4. History of alcohol or narcotic drug abuse, or a history of mental illness, confrontational personality, bad motivation, paranoia, or other emotional or intellectual problems that may affect the informed validity of participation in this study
5. Preoperative respiratory infection, allergic rhinitis, bronchial asthma, chronic obstructive pulmonary disease, postnasal drip syndrome, oral ACEI drugs, CVA, EB, obvious acid reflux, heartburn, etc.
6. Patients with severe cardiac insufficiency or heart-related diseases before surgery
7. Diabetes before surgery
8. Severe liver and kidney damage before surgery

8) ACEI/ARB used within 1 month 9) Use of drugs that may cause cough or suppress cough within 1 month 9) Preoperative narrow-angle glaucoma, benign prostatic hyperplasia, or bladder neck obstruction 10) Patients who are using beta2 agonists or acetylcholine receptor antagonists or inhaled glucocorticoids 11) Tumor recurrence 13) Patients with severe infection or obvious pleural effusion found on postoperative chest X-ray

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of significant cough two weeks after surgery | 12 weeks
  Cough Evaluation Test (CET) is an easy way to assess the cough condition. A Visual Analogue Scale (VAS) is a cough rating scale. Significnant cough means VAS more than 3 or any item of CET score more than 2.

SECONDARY OUTCOMES:
The total and sub-scores of the Cough Evaluation Test (CET) score of each day after surgery | 12 weeks
  Cough Evaluation Test (CET) is an easy way to assess the cough condition
Incidence of significant cough 1 month after surgery | 12 weeks
  Cough Evaluation Test (CET) is an easy way to assess the cough condition. A Visual Analogue Scale (VAS) is a cough rating scale. Significnant cough means VAS more than 3 or any item of CET score more than 2.
LCQ-MC at 1 month after surgery | 12 weeks
  Leicester Cough Questionnaire in Mandarin-Chinese (LCQ-MC) is a useful questionnaire to evaluate cough after surgery
the number of days the cough lasts | 12 weeks
  the number of days the cough lasts
Cough start time | 12 weeks
  Days from surgery to onset of cough
Inflammatory factor levels in venous blood before and after surgery | 12 weeks
  we test the inflammatory factor 3 days before surgery and 1 day after surgery
Incidence of serious postoperative pneumonia | 12 weeks
  we make a chest radiograph after surgery to find the postoperative pneumonia
length of postoperative hospital stay | 12 weeks
  length of postoperative hospital stay

REFERENCES:
- [Derived] Dong J, Jiang S, Qiu Y, Li J, Cui F, Liang H, Lao S, Xie Z, Huang J, Hao Z, He H, Xv X, Zhang M, He M, Zhang Y, He J, Wang W. Budesonide/glycopyrronium/formoterol fumarate co-suspension metered dose inhaler relieves cough after lobectomy: a randomized controlled study. Transl Lung Cancer Res. 2025 Apr 30;14(4):1290-1300. doi: 10.21037/tlcr-24-905. Epub 2025 Apr 27. PMID 40386713